CLINICAL TRIAL: NCT04759352
Title: Cancer Genetic Counseling: Telephone Versus Standard In-person Delivery. A Randomized Trial (GEO-STAR)
Brief Title: Telephone Versus In-person Post-test Cancer Genetic Counseling
Acronym: GEO-STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Daniela Turchetti, Prof., IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GEO-STAR
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cancer Gene Mutation
Keywords: genetic telecounselling; test result communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone post-test genetic counseling (Experimental): Post-test genetic counseling delivered by telephone
  Interventions: Other: Post-test genetic counseling delivered by telephone
- In-person post-test genetic counseling (No Intervention): Post-test genetic counseling delivered in-person

INTERVENTIONS:
Other: Post-test genetic counseling delivered by telephone — Participants enrolled in the experimental arm will receive genetic counseling for test result communication by telephone.
  Arms: Telephone post-test genetic counseling

SUMMARY:
The purpose of the GEO-STAR randomized non-inferiority trial is to compare the outcome of post-test telephone cancer genetic counseling with standard in-person cancer genetic counseling. We hypothesize that telephone counseling is non-inferior by outcome if compared to standard in-person counseling.

DETAILED DESCRIPTION:
Consecutive patients undergoing pre-test cancer genetic counseling and cancer genetic testing, during the study period, will be eligible to participate. During the pre-test genetic counseling, demographic data, family and personal medical history will be collected and pedigree will be drawn. Available participants will provide written informed consent. They will be then randomized in blocks of ten participants using an online system (http://wwwservizi.regione.emilia-romagna.it/generatore/).

The study is open label; thus, patients and investigators will not be blinded to treatment allocation due to the study nature intervention.

After randomization, participants will be scheduled for post-test genetic counseling session. Participants randomized to usual care will receive standard in-person result disclosure. Participants randomized to telephone counseling will be scheduled for telephone post-test counseling sessions. One-week after completing the post-test genetic counseling session, the survey package will be sent by email to participants to assess impact and satisfaction with post-test counseling.

Genetic counselors delivering post-test genetic counseling will complete the questionnaire immediately after the post-test session.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age inclusive at the time of the study;
* Patients must have undergone an in-person pre-test genetic counseling session;
* Patients must have undertaken cancer genetic testing;
* Patients must be able to speak Italian fluently;
* Patients must have got an email address.

Exclusion Criteria:

* Patients unable to provide informed consent, for example due to mental incapacity or active psychotic illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
"Multidimensional Impact of Cancer Risk Assessment" questionnaire | Seven days after the post-test genetic counseling session
  Impact of post-test counseling on patients. The "Multidimensional Impact of Cancer Risk Assessment" questionnaire measures distress, uncertainty and positive experiences associated to cancer genetic testing. A version adapted to the Italian context will be used, where a single item related to insurance has been removed because not applicable to the Italian Health System. The resulting possible scores range from 0 to 100. Higher scores indicate more negative impacts of cancer risk assessment.
"Patient perceptions of the genetic counseling questionnaire" | Seven days after the post-test genetic counseling session
  Impact of post-test counseling on patients. The range of scores is from 8 to 31. Higher scores indicate positive perception of the genetic counseling session.
"Genetic Counselor process Questionnaire" | Immediately after the post-test genetic counseling session
  Professionals perceptions measured by the Genetic Counselor process Questionnaire completed by professionals who provided the post-test genetic counseling. The range of scores is from 4 to 20. Higher scores indicate positive perception of the genetic counselor.

SECONDARY OUTCOMES:
Influence of sociodemographic and medical history on genetic counseling outcomes | Data collection during pre-test genetic counseling session
  Sociodemographic variables and family and personal cancer history will be collected during the pre-test session.
Impact of logistics on genetic counseling preferences | Data collection during the pre-test genetic counseling session
  Distance (in kilometers) of patient's primary residence to the clinic location collected by the demographic data collected at pre-test genetic counseling

CONTACTS AND LOCATIONS:
Locations (1):
- UO Genetica Medica, IRCCS AOU di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No